CLINICAL TRIAL: NCT03413605
Title: A Multilevel CBPR Intervention to Improve Colorectal Cancer Screening in Underserved Vietnamese Americans
Brief Title: U01 CRC Project for Vietnamese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U01 Viet CRC; U01MD010627 (NIH)
Record Dates: First submitted 2017-12-11; First posted 2018-01-29 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a multilevel CBPR intervention (Experimental): The intervention will be delivered in group-based education workshop format. The education session is a curriculum-based group education; each group will be having about 15-20 participants. We will allow 5-7 minutes for participants to get to know each other and to get comfortable talking to the group. Education will have two major topics.(a) CDC's standard Clinical Preventive Services Guidelines for adults 50+ (CPS). (b) culturally tailored CRC information discussion. This session is to increase knowledge, change cultural beliefs and attitudes on risks of CRC and benefits of screening by using interactive discussion approaches, visual aids, motivation video and print materials.
  Interventions: Behavioral: A Multilevel CBPR Intervention
- control group (No Intervention): the standard CDC's Clinical Preventive Services Guidelines for adults 50+ (CPS) will be provided to control groups.

INTERVENTIONS:
Behavioral: A Multilevel CBPR Intervention — The intervention will be implemented through a group-based education workshop. The education session is a curriculum-based group education; each group will be having about 15-20 participants. All group education sessions will take place at collaborating Viet community partners sites, and delivered in Vietnamese language, with offering of refreshment. We will allow 5-7 minutes for participants to get to know each other and to get comfortable talking to the group. Education will have two major topics--- (a) CDC's standard Clinical Preventive Services Guidelines for adults 50+ (CPS). (b) culturally tailored CRC information discussion.
  Arms: a multilevel CBPR intervention

SUMMARY:
Colorectal cancer (CRC) is the second most commonly diagnosed cancer and the third highest cause of mortality in Vietnamese and Asian Americans. CRC incidence is rising rapidly in Vietnamese Americans, but they have among the lowest rates of CRC screening (14%) and are more likely to be diagnosed with advanced stage disease, which is highly preventable. Over 85% of Vietnamese Americans in our region (PA, NJ and NYC) are foreign-born with limited English proficiency, have low SES, and live in economically disadvantaged neighborhoods. Many lack knowledge about CRC risks and screening benefits and have limited access to culturally appropriate preventive care. Center for Asian Health, Temple University will be working with Vietnamese CBOs to address their critical health disparities. The investigators will test the hypothesis that the proposed multilevel CRC intervention will yield higher CRC screening rates compared to the control at 12-month follow-up. This project represents the first large-scale community-based randomized controlled trial of a multilevel, culturally-appropriate intervention to increase CRC screening among underserved Vietnamese. If effective, this innovative CRC intervention can be used as a model program that has potential impact, generalizability and sustainability in Asian American and other underserved ethnic communities.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most commonly diagnosed cancer and the third highest cause of mortality in Vietnamese and Asian Americans. CRC incidence is rising rapidly in Vietnamese Americans, but they have among the lowest rates of CRC screening (14%) and are more likely to be diagnosed with advanced stage disease, which is highly preventable. Over 85% of Vietnamese Americans in our region (PA, NJ, and NYC) are foreign-born with limited English proficiency, have low SES, and live in economically disadvantaged neighborhoods. Many lack knowledge about CRC risks and screening benefits and have limited access to culturally appropriate preventive care. Thus, a multilevel intervention is needed to address the multiple barriers to and determinants of CRC screening in this community. Vietnamese community organizations (VCOs) serve dynamic social functions and represent an important resource for addressing this critical health disparity priority by promoting CRC screening. This project builds on established partnerships and successful work of Center for Asian Health, Temple University with Vietnamese CBOs that address their overwhelming health disparities. CBPR principles will be applied to engage 20 VCOs in all phases of planning, implementing, evaluating, and disseminating a culturally appropriate, theory- and evidence-based multilevel CRC intervention. The proposed intervention will be guided by Social Ecological Model, which addresses sociocultural, behavioral and environmental determinants and intervention strategies at the individual, interpersonal, and community organizational levels. CDC's Clinical Preventive Services Guidelines for adults 50+ (CPS) recommend that cancer screenings and other preventive services should be promoted. The standard CPS will be provided to both intervention and control groups, and intervention group will receive CPS + multilevel CRC intervention. Specific Aim 1 is to test the hypothesis that CPS + multilevel CRC intervention will yield higher CRC screening rates compared to CPS control at 12-month follow up; Aim 2 is to examine whether CPS + multilevel CRC intervention (which includes CHW-led group education, automated and interactive text messaging and phone-based peer support) is more effective in changing screening determinants (e.g. KAB, self-efficacy, risk factors, lifestyles, social support, social norms, access barriers) than CPS control condition; and Aim 3 is to assess costs and cost-effectiveness of CPS + multilevel CRC intervention compared to CPS control condition in relation to CRC screening rates in order to inform future dissemination efforts. In sum, this project represents the first large-scale community-based randomized controlled trial of a multilevel, culturally-appropriate CBPR intervention to increase CRC screening among underserved Vietnamese. If effective, this innovative multilevel CRC intervention can be used as a model program that has potential generalizability and sustainability in Asian American and other underserved ethnic communities to impact preventive behaviors at the population level.

ELIGIBILITY:
Inclusion Criteria:

1. self-identified Vietnamese ethnicity,
2. age 50 and above,
3. accessible by cell telephone,
4. presence in the same geographic study area for a period of one year (to minimize participant attrition);
5. not enrolled in any CRC intervention (to prevent a potential program impact),
6. do not have the colorectal polyp, CRC cancer or a family history of CRC (first-degree relative),
7. non-adherent to CRC screening guidelines (never had CRC screening or are overdue for screening).

Exclusion Criteria:

1. enrolled in any CRC intervention (to prevent a potential program impact)
2. have the colorectal polyp, CRC cancer or a family history of CRC
3. had CRC screening or adherent to CRC screening guidelines

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace X Ma, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Vietnamese community center of Atlantic city, Atlantic City, New Jersey
  - Bo De Temple, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- a Multilevel CBPR Intervention: The intervention was delivered in group-based education workshop format. The education session was a curriculum-based group education; each group had about 15-20 participants. We allowed 5-7 minutes for participants to get to know each other and to get comfortable talking to the group. Education had two major topics.(a) CDC's standard Clinical Preventive Services Guidelines for adults 50+ (CPS). (b) culturally tailored CRC information discussion. This session was aimed to increase knowledge, change cultural beliefs and attitudes on risks of CRC and benefits of screening by using interactive discussion approaches, visual aids, motivation video and print materials.
- Control Group: the standard CDC's Clinical Preventive Services Guidelines for adults 50+ (CPS) was provided to control groups.
Period: Overall Study Baseline
Arm/Group | a Multilevel CBPR Intervention | Control Group
Started | 392 | 409
Completed | 392 | 409
Not Completed | 0 | 0
Period: Post Intervention Assessment
Arm/Group | a Multilevel CBPR Intervention | Control Group
Started | 392 | 409
Completed | 392 | 409
Not Completed | 0 | 0
Period: 12-m Follow up
Arm/Group | a Multilevel CBPR Intervention | Control Group
Started | 392 | 409
Completed | 364 | 382
Not Completed | 28 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | a Multilevel CBPR Intervention | Control Group | Total
Number analyzed (Participants) | 392 | 409 | 801
Age, Customized [Count of Participants; unit: Participants]
  50-74 years old | 325 | 321 | 646
  75 or older | 67 | 88 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 252 | 474
  Male | 170 | 157 | 327
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Nativity Status [Count of Participants; unit: Participants] — Population: n=13 participants did not report their nativity status.
  Participants
    Foreign Born: number analyzed (Participants) | 386 | 402 | 788
    Foreign Born | 384 | 399 | 783
    US Born: number analyzed (Participants) | 386 | 402 | 788
    US Born | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Screening Rate
Description: percentage of subjects, who received colorectal screening at 12-month Follow Up
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | a Multilevel CBPR Intervention | Control Group
Number analyzed (Participants) | 364 | 382
Participants | 333 | 162

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | a Multilevel CBPR Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/392 | 0/409
Serious Adverse Events (participants affected / at risk) | 0/392 | 0/409
Other Adverse Events (participants affected / at risk) | 0/392 | 0/409

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03413605/Prot_SAP_000.pdf